## Statistic analysis

The data will be expressed as a mean  $\pm$  SD. For continuous variables, the variations between the groups are compared by means of the averages calculated with the non parametric Wilcoxon and Mann-Whitney U tests. The variability of the biochemical parameters over time will be evaluated by means of tests for repeated measurements. A correlation analysis will be performed with the Pearson correlation test, after adequate logarithmic transformation of the parameters when necessary. Multiple regression analysis will be used to evaluate associations between variables. Statistical significance will be assumed for values of p <0.05. All statistical analyzes will be performed with the SPSS program for Windows version 22.0 (SPSS INC; Chicago, IL, USA).

All children with T1D with disease onset in the years 2017, will receive omega 3 supplement (EPA + DHA 60 mg / kg / of), and will be compared from a metabolic point of view (in particular for the needs of insulin and glycated hemoglobin) according to the scheme outlined with the pre-supplementation data, deduced from the medical records retrospectively.

## supplementation omega-3 $\downarrow$

| Group 1 n. | Group 2 n. | Group 3 n. | Group 4 new onset | |
|------------|------------|------------|-------------------|------|
| | vs Group 1 | vs Group 2 | vs Group 3 | |
| | | vs Group 1 | vs Group 2 | |
| | | | vs Group 1 | |
| 2014 | 2015 | 2016 | 2017 | 2018 |

The analysis will allow to quantify the effects of omega-3 at different distance from the onset in terms of metabolic advantage (insulin units / Kg / die, glycated hemoglobin, etc.) and to evaluate if and how much supplementation after the onset may give metabolic advantages compared to other patients not yet supplemented.

Further statistical analysis could be performed if appropriate.